CLINICAL TRIAL: NCT00193531
Title: Phase II Study of Paclitaxel, Carboplatin, and Oral Etoposide Followed by Weekly Paclitaxel in the Treatment of High Grade Neuroendocrine Carcinoma
Brief Title: Paclitaxel, Carboplatin, and Oral Etoposide Followed by Weekly Paclitaxel in High Grade Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MISC 16
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Paclitaxel; Carboplatin; Etoposide

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin
Drug: Etoposide

SUMMARY:
carboplatin and etoposide, followed by maintenance therapy with weekly paclitaxel in patients with poorly differentiated neuroendocrine carcinomas. We hope to identify a "standard treatment" for this unusual group of patients who are not usually eligible for clinical trials.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Paclitaxel + Carboplatin + Etoposide

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic poorly differentiated neuroendocrine carcinoma
* Unknown primary site
* Able to perform activities of daily living with minimal assistance
* Measurable or evaluable disease
* Adequate bone marrow, liver functions and kidney function
* No previous treatment with chemotherapy
* Understand the nature of this study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* Previous malignancy within five years
* Women pregnant or lactating
* Recent history of cardiovascular disease
* Meningeal metastases

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1998-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall response

SECONDARY OUTCOMES:
Overall survival
Time to progression
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Litchy S, Greco FA. Phase II trial of paclitaxel, carboplatin, and etoposide in advanced poorly differentiated neuroendocrine carcinoma: a Minnie Pearl Cancer Research Network Study. J Clin Oncol. 2006 Aug 1;24(22):3548-54. doi: 10.1200/JCO.2005.05.0575. PMID 16877720